CLINICAL TRIAL: NCT01870193
Title: Glutathione and Fuel Oxidation in Aging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rajagopal V Sekhar (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Rajagopal V Sekhar, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: H-30681 GSH-Aging; R01AG041782 (NIH)
Record Dates: First submitted 2013-05-30; First posted 2013-06-05 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Aging
Keywords: Glutathione deficiency in aging; Impaired mitochondrial fatty-acid oxidation in aging
MeSH Terms: interventions — Glycine; Cysteine; Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Young controls (Active Comparator): Young controls will be studied before and after receiving cysteine and glycine for 2 weeks
  Interventions: Dietary Supplement: Glycine, cysteine (as n-acetylcysteine), alanine
- Elderly active (Active Comparator): Elderly subjects in the active group will receive glycine plus cysteine (as n-acetylcysteine) for 4 months, and be studied at baseline, 2 weeks and 4 months
  Interventions: Dietary Supplement: Glycine, cysteine (as n-acetylcysteine), alanine
- Elderly placebo (Placebo Comparator): Elderly subjects in the placebo group will receive alanine for 4 months, and be studied at baseline, 2 weeks and 4 months
  Interventions: Dietary Supplement: Glycine, cysteine (as n-acetylcysteine), alanine

INTERVENTIONS:
Dietary Supplement: Glycine, cysteine (as n-acetylcysteine), alanine — Young controls will receive cysteine plus glycine for 2 weeks
  The elderly subjects will be randomized in a double-blinded design to receive either cysteine plus glycine OR alanine for a period of 4 months

SUMMARY:
Glutathione is an important antioxidant protein which protects cells from harmful oxidative stress. Elderly humans are known to have elevated oxidative stress and deficiency of glutathione, but it is not known whether there is deficient synthesis of glutathione in muscle tissue of elderly humans.

Mitochondria are engines of cells where food consumed is burned to make energy. Under normal conditions the fuel of choice in the fasted state is fat, but fasted elderly humans are not able to oxidize fat as well as healthy young humans. Elderly humans also have the highest incidence and prevalence of being overweight and obese, and have increased storage of fat in liver and muscle.

This study will help determine whether

1. elderly humans have diminished synthesis of glutathione in the skeletal muscle, and whether this can be improved by supplementing cysteine and glycine (and not an isonitrogenous placebo) in the diet;
2. improving muscle glutathione concentrations can also improve fuel oxidation in aging;
3. improvement of intracellular glutathione concentrations will be associated with a change in total body fat content

DETAILED DESCRIPTION:
Subjects will be recruited by written informed consent on forms approved by the Institutional Review Board of Baylor College of Medicine at the time of approval of the full protocol. Subjects taking an nonvitamin supplements or lipid lowering medications will stop this 4 weeks before the screening labs and for the entire duration of the study. Fasted subjects will have screening labs (blood count, HbA1c, lipid profile, liver profile, blood urea nitrogen, Creatinine, thyroid stimulating hormone, free t4, cortisol) followed by an oral glucose tolerance test, measures of muscle strength by dynamometry, tests of function (including a 6-min walk test) and body composition scans to measure total body fat. On another occasion, fasted subjects will be undergo stable isotope infusions and other studies in the metabolic research unit to measure concentrations of amino-acids and glutathione in red blood cells and muscle tissue, glutathione synthesis rates in muscle and red cells, plasma and whole-body mitochondrial fatty-acid oxidation, Kreb's cycle function, urine urea nitrogen, plasma reactive oxygen species and F2-isoprostanes, genes of glutathione synthesis and fuel oxidation. Elderly subjects will also have magnetic resonance spectroscopy scan for liver and muscle fat content.

Young subjects will be given dietary cysteine and glycine for 2-weeks and be restudied 2-weeks later. They are then released from the study.

Elderly subjects will be studied for 16 weeks. They will be assigned to receive either cysteine plus glycine, or alanine in a randomized, double-blinded study design. The studies described above will be repeated after 2 weeks and 16 weeks. Subjects will have monthly measures of liver profile, lipid profiles, BUN and creatinine and glutathione.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly subjects: age range 61-80y.
2. Young healthy subjects: age range 21-40y

Exclusion Criteria:

1. Renal impairment (serum creatinine >1.5 mg/dL)
2. Liver impairment (liver transaminases >2x upper limit of normal)
3. Untreated/uncontrolled hyperthyroidism or hypothyroidism
4. Known hypercortisolemia
5. Known diabetes mellitus
6. Hospitalization in the past 3 months
7. BMI <27 (elderly group)
8. Elderly women on estrogen replacement
9. Known pre-existing coronary artery disease
10. Fasted plasma triglyceride >300 mg/dl (on lipid lowering medications)
11. Fasted plasma triglyceride >500 mg/dl (off lipid lowering medications)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-04-23 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Muscle glutathione concentration | Each subject will be studied over 4 months

CONTACTS AND LOCATIONS:
Overall Officials: R V Sekhar, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar P, Liu C, Suliburk J, Hsu JW, Muthupillai R, Jahoor F, Minard CG, Taffet GE, Sekhar RV. Supplementing Glycine and N-Acetylcysteine (GlyNAC) in Older Adults Improves Glutathione Deficiency, Oxidative Stress, Mitochondrial Dysfunction, Inflammation, Physical Function, and Aging Hallmarks: A Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2023 Jan 26;78(1):75-89. doi: 10.1093/gerona/glac135. PMID 35975308